CLINICAL TRIAL: NCT02180802
Title: Parental Involvement Improves the Effect of Motivational Interviewing on Weight Loss in Obese Adolescents: A Randomized Controlled Trial Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qazvin University Of Medical Sciences (Other)
Responsible Party: Principal Investigator, Amir H Pakpour, vice dean for research, Qazvin University Of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 3287
Record Dates: First submitted 2014-07-01; First posted 2014-07-03 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-08

CONDITIONS: Obesity, Adolescent
Keywords: obese adolescents; BMI ≥ 95th percentile for age and gender
MeSH Terms: conditions — Pediatric Obesity; Coitus | interventions — Motivational Interviewing; Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- motivational intervieing group (Experimental): The behavioral intervention targets were improved eating and physical activity behavior in order to reduce obesity levels. Each adolescent was encouraged to eat a variety of foods from each of the four major food groups and low-fat alternatives . Moreover, each adolescent was encouraged to achieve at least 60 minutes of moderate-to-vigorous intensity physical activity daily as recommended by the World Health Organization
  Interventions: Behavioral: motivational interviewing
- motivational interviewi group with parental involvement (Experimental): an additional single session with parents or guardians over 60 minutes in the clinic
  Interventions: Behavioral: motivational interviewing with parental involvement
- Control (Active Comparator): The patients received routine care
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: motivational interviewing
  Arms: motivational intervieing group
Behavioral: motivational interviewing with parental involvement
  Arms: motivational interviewi group with parental involvement
Behavioral: Control group
  Arms: Control

SUMMARY:
Motivational interviewing (MI) has been shown to be an effective strategy in targeting obesity in adolescents and parental involvement has been associated with increased effectiveness. The aim of the study is to evaluate and compare the role of parental involvement in MI interventions for obese adolescents

ELIGIBILITY:
Inclusion Criteria:

* BMI equal or higher than 95th percentile for age and gender
* 13-18 years old

Exclusion Criteria:

* medication with weight gain as side effects
* diagnosed with having eating disorder
* pregnant
* clinical mental health conditions
* psychosis

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 408 (Actual)
Dates: Start 2011-02; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
changes in BMI | changes from baseline and 12 months follow-up
  Body Mass Index
Child Dietary Self-Efficacy | changes from baseline and 12 months follow-up
  Child Dietary Self-Efficacy Scale (CDSS)
Weight Efficacy Lifestyle | changes from baseline and 12 months follow-up
  Weight Efficacy Lifestyle questionnaire (WEL)
Physical Exercise Self-efficacy | changes from baseline and 12 months follow-up
  Physical Exercise Self-efficacy Scale (PES)
changes in physical activity | changes from baseline and 12 months follow-up
changes in dietary pattern | changes from baseline and 12 months follow-up

SECONDARY OUTCOMES:
Changes in blood cholesterol level | changes from baseline and 12 months follow-up
changes in blood triglyceride level | changes from baseline and 12 months follow-up
Changes in body fat percentage | changes from baseline and 12 months follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Pediatric Clinic, Qazvin, Qazvin Province, Iran